CLINICAL TRIAL: NCT04299659
Title: Comparison of Four Methods for Entering the Gap Position of Landolt Cs With Respect to Validity, Retest Reliability, Examination Duration and Test Subject Satisfaction
Brief Title: Comparison of Four Methods for Entering the Gap Position of Landolt Cs
Acronym: LC_Entry
Status: Completed | Type: Observational
Sponsor: Aalen University (Other)
Responsible Party: Sponsor
Other Study IDs: LC Entry_2020
Record Dates: First submitted 2020-03-01; First posted 2020-03-09 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Quality Control; Validation Study
Keywords: psychophysics; visual acuity; response; response entry; validity; retest reliability; reproducibility; evaluation; optotype; Landolt C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Landolt C entry method — Four different methods for entering the Landolt C gap position are compared

SUMMARY:
The aim of this study is to investigate and compare the validity of four different input methods for Landolt Cs, i.e. the proportion of correct gap positions in relation to the total number of performances. The four input methods are a numeric keypad, an eight-positions rocker switch, a remote control and voice feedback.

DETAILED DESCRIPTION:
The measurement of visual acuity is the most frequent and one of the most important ophthalmological functional investigations. Therefore, it is particularly important to find a measuring procedure with as little input errors as possible.

The 8-position Landolt C (LC) is the internationally accepted, well-standardised optotype for the determination of visual acuity.

Usually, the subjects informs the examiner verbally about the perceived position of each LC. According to the current literature, about 20 to 30 % of the population suffers from a right/left weakness. Furthermore, language barriers are an additional considerable hurdle.

Therefore, it is important to find an input method for the LC gap positions with minimal entry mistakes. In oder to avoid the thresholding procedure and its inherent difficulties, highly supra-threshold (10 times above the previously determined individual central visual acuity threshold) 8-position LCs are presented.

The study compares four input methods for entering of the Landolt C gap positions: a modified numeric keypad, an 8-position rocker switch, a modified TV remote control and voice/verbal feedback.

Each subject will perform all four input methods, with 2 test runs of 16 Landolt C presentations, each. A forced-choice method will be applied, i.e. the test is not continued until the test person has responded ot each single presentation. Regardless of whether the entry was correct or incorrect, the next Landolt C is displayed.

The optotypes are presented using modified version of the Freiburg Visual Acuity and Contrast Test (FrACT), which allows to present the 8-position Landolt Cs in a standardized way on a video display unit (VDU).

The sequence of the input methods is randomized. This study is carried out in a "within-subject design", i.e. all test persons go through all test conditions and serve as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Informed consent
* (Distance) visual acuity with best correction: ≥ 0.8
* (Distant) ametropia: ≤+8.0 Diopters (spherical equivalent)
* Anisometropia ≤ 3 dpt
* Astigmatism ≤ 2.5 dpt

Exclusion Criteria:

* Prolonged reaction time caused by drugs (medications)/ drugs/alcohol
* Movement disorders (of hands) such as Parkinson's disease
* Indication of amblyopia (strabismus surgery, occlusion therapy etc.)
* Eye movement disorders/double vision
* Defective stereo vision (according to LANG [I] stereo test)
* Presence of a relative afferent pupil defect ("swinging flashlight test)
* Any hint of visual pathway lesion or other chronic or progressive eye disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, young subjects recruited for the students and or co-workers of the Aalen University of Applied Sciences
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
validity | Through study completion, an average of 3 months
  Proportion of correct gap position entries in relation to the total number of LC presentations by the four different entry methods

SECONDARY OUTCOMES:
retest reliability | Through study completion, an average of 3 months
  Comparison of the correct gap position entry between first and second test run by the four different entry methods
Examination duration | Through study completion, an average of 3 months
  Comparison of the examination duration of the the four different entry methods and by the first and second run
Subjects´ satisfaction | Through study completion, an average of 3 months
  Subjects´ evaluation (using a questionnaire) for the four different entry methods

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, M.D., Study Chair — +49 7361 576-4605
Locations (1):
- Ulrich SCHIEFER, Aalen, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No